CLINICAL TRIAL: NCT06262217
Title: Mobile MRI for Immediate Radiological Acute Cerebral Lesion Evaluation in Stroke: Investigating the Use of a Small Mobile MRI Scanner to Aid Investigation of Stroke
Brief Title: Mobile MRI for Immediate Radiological Acute Cerebral Lesion Evaluation in Stroke
Acronym: MIRACLES
Status: Recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: INGN21ST510
Record Dates: First submitted 2023-03-27; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Mobile MRI: Mobile MRI scan
  Interventions: Device: Mobile MRI scanner

INTERVENTIONS:
Device: Mobile MRI scanner — Use of mobile MRI scanner in patients with suspected or confirmed acute stroke (including Transient Ischaemic attacks)

SUMMARY:
This prospective observational study will evaluate the potential value of mobile MRI in patients with suspected or proven acute stroke and Transient Ischemic Attack (TIA), undertaking additional imaging in the emergency department, acute stroke unit, or outpatient settings, and comparing diagnostic accuracy, Diffusion-weighted imaging (DWI) lesion volume and detection of complications (brain swelling or haemorrhagic transformation). Information on ease of use, tolerability and image quality will also be gathered.

DETAILED DESCRIPTION:
The study will investigate mobile MRI for immediate radiological acute cerebral lesion evaluation in Stroke. The objectives are:

1. Among patients with possible acute minor stroke or TIA, to compare the detection rate of acute DWI lesions on mobile MRI scan with routine imaging, describe number and distribution of lesions, and describe the intervals between mobile MRI and routine diagnostic scan, and time to final clinical diagnosis
2. Among patients with acute stroke of uncertain onset time, to compare the presence of DWI-Fluid attenuated inversion recovery (FLAIR) mismatch pattern on mobile MRI with CT perfusion (CTP) mismatch.
3. Among patients with confirmed acute ischaemic stroke, to compare the volume of DWI lesion on mobile MRI with the core volume on CTP
4. Among patients with established stroke post-thrombolysis or thrombectomy, to compare the incidence of brain swelling and haemorrhagic transformation on mobile MRI with routine imaging
5. In all groups, to evaluate the tolerability and ease of use of the mobile MRI scanner, and to rate image quality

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female > or = 18 years of age
* Clinically suspected stroke or transient ischaemic attack, or confirmed clinical diagnosis of stroke or TIA
* Consent of patient or legal representative

Exclusion Criteria:

* Contraindications to MRI brain scan as per standard MRI checklist for NHS Greater Glasgow & Clyde

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically suspected stroke or transient ischaemic attack, or confirmed clinical diagnosis of stroke or TIA
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic sensitivity and specificity of mobile MRI scanner | 1 week
  In patients with suspected or confirmed acute stroke (including transient ischaemic attack), what is the sensitivity and specificity of scans obtained with a mobile low field MRI scanner compared to routine diagnostic scanning

SECONDARY OUTCOMES:
Comparison of MRI abnormalities | 1 week
  Number, size and location of mobile MRI abnormalities compared to routine scanning with MRI or CT (including CT perfusion scans to examine brain blood flow)
Final Clinical Diagnosis | 3 months
  Final clinical diagnosis and level of confidence in diagnosis
Final Clinical Diagnosis | 3 months
  Final clinical diagnosis
Time from arrival at the Emergency Department to scan | 2 weeks
  Time from hospital arrival to scan in acute patients
Use of treatments | 3 months
  Use of treatments (acute or to deal with complications of stroke)
Patient Outcomes | 3 months
  Disability at 3 months after stroke using modified rankin scale with higher scores corresponding to worse outcomes
Level of confidence in final diagnosis | 3 months
  Level of confidence in final diagnosis on scale of possible, probable or definite

CONTACTS AND LOCATIONS:
Overall Officials: Keith W Muir, MD, Principal Investigator — University of Glasgow
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No